CLINICAL TRIAL: NCT02237729
Title: Phase 1, Double Blind, Randomized, Parallel-group, 3-arm, Single-dose, Comparative Pharmacokinetic Study Of Pf-06410293 and Adalimumab Sourced From Us And Eu Administered To Healthy Male And Female Subjects
Brief Title: A Study Of PF-06410293 (Adalimumab-Pfizer) And Adalimumab (Humira) In Healthy Subjects (REFLECTIONS B538-07))
Acronym: B538-07
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: B5381007; REFLECTIONS B538-07
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Healthy Subjects
Keywords: healthy subjects; immunology; PK; Phase 1; bioequivalence; biosimilarity; adalimumab; single dose.
MeSH Terms: interventions — PF-06410293

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PF-06410293 (Experimental)
  Interventions: Biological: PF-06410293
- Adalimumab-US (Active Comparator)
  Interventions: Biological: Adalimumab-US
- Adalimumab-EU (Active Comparator): Adalimumab-EU will be administered as a single 40 mg, subcutaneous dose
  Interventions: Biological: Adalimumab-EU

INTERVENTIONS:
Biological: PF-06410293 — PF-06410293 will be administered as a single 40 mg, subcutaneous dose
  Other Names: Adalimumab-Pfizer
  Arms: PF-06410293
Biological: Adalimumab-US — Adalimumab-US will be administered as a single 40 mg, subcutaneous dose
  Arms: Adalimumab-US
Biological: Adalimumab-EU — Adalimumab-EU will be administered as a single 40 mg, subcutaneous dose
  Arms: Adalimumab-EU

SUMMARY:
This is a Phase 1, double blind (sponsor open), randomized (1:1:1), parallel group, 3 arm, single dose comparative PK study of adalimumab Pfizer and adalimumab sourced from the US and EU administered subcutaneously (SC) to healthy male and female volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects between the ages of 18 and 45 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, complete physical examination including blood pressure and heart rate measurement, 12 lead ECG and clinical laboratory tests.
* Body Mass Index (BMI) of 19.0 to 30.5 kg/m2; and a total body weight >60 kg (132 lbs).
* Chest X ray with no evidence of current, active TB or previous (inactive) TB, general infections, heart failure, malignancy, or other clinically significant abnormalities taken at Screening or within 24 weeks prior to Day 1 and read by a qualified radiologist.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, autoimmune, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Previous history of cancer, except for adequately treated basal cell or squamous cell carcinoma of the skin.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 362 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
maximal serum concentration (Cmax) | Day 1 - Day 50
  maximal serum concentration (Cmax)
area under the concentration time curve (AUC) from time 0 to 2 weeks (AUC0-2wk) | 0-336 hours
  area under the concentration time curve (AUC) from time 0 to 336 hours (AUC0-2wk)
Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-T)] | Day 1 - Day 50
  AUC (0-T)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-T)
AUC extrapolated to infinity (AUC0inf) | Day 1 - Day 50
  AUC extrapolated to infinity (AUC0inf)

SECONDARY OUTCOMES:
Type, incidence, severity, timing, seriousness and relatedness of treatment emergent adverse events, and abnormalities in laboratory parameters | Day 1- Day 71
  Type, incidence, severity, timing, seriousness and relatedness of treatment emergent adverse events, and abnormalities in laboratory parameters
Incidence of antidrug antibodies (ADA) and neutralizing antibodies (NAb) | Day 1- Day 71
  Incidence of antidrug antibodies (ADA) and neutralizing antibodies (NAb)
maximal serum concentration (Cmax) for adalimumab EU as compared to adalimumab US | Day 1 - Day 50
  maximal serum concentration (Cmax) for adalimumab EU as compared to adalimumab US
area under the concentration time curve (AUC) from time 0 to 2 weeks (AUC0-2wk) for adalimumab EU as compared to adalimumab US | 0-336 hours
  area under the concentration time curve (AUC) from time 0 to 336 hours (AUC0-2wk) for adalimumab EU as compared to adalimumab US
Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-T)] for adalimumab EU as compared to adalimumab US | Day 1 - Day 50
  AUC (0-T)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-T) for adalimumab EU as compared to adalimumab US
AUC extrapolated to infinity (AUC0inf) for adalimumab EU as compared to adalimumab US | Day 1 - Day 50
  AUC extrapolated to infinity (AUC0inf) for adalimumab EU as compared to adalimumab US
time to reach the maximum concentration (Tmax) | Day 1 - Day 50
  time to reach the maximum concentration (Tmax)
Apparent clearance (CL/F) | Day 1 - Day 50
  Apparent clearance (CL/F)
Apparent volume of distribution (Vz/F) | Day 1 - Day 50
  Apparent volume of distribution (Vz/F)
Terminal half-life (T1/2) | Day 1 - Day 50
  Terminal half-life (T1/2)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (7):
  - De La Pedraja Radiology Associates, Coral Gables, Florida
  - SeaView Jacksonville, Jacksonville, Florida
  - SeaView Research, Inc., Miami, Florida
  - SeaView Reseach Screening Office, Miami, Florida
  - SeaView Research, Inc. (Screening Office), Miami, Florida
  - Vince & Associates Clinical Research, Inc., Overland Park, Kansas
  - Prism Research, LLC, Saint Paul, Minnesota

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5381007&StudyName=A%20Study%20Of%20PF-06410293%20%28Adalimumab-Pfizer%29%20And%20Adalimumab%20%28Humira%29%20In%20Healthy%20Subjects%20%28REFLECTIONS%20B538-07%29%29